CLINICAL TRIAL: NCT05773586
Title: A Phase 1 Study to Evaluate Safety and Tolerability, Pharmacokinetics and Preliminary of APG-5918 in Healthy Subjects or Anemic Patients
Brief Title: A Study to Investigate the Safety, Pharmacokinetics and Efficacy of APG-5918 in Healthy Subjects or Anemic Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APG5918AC101
Record Dates: First submitted 2023-02-22; First posted 2023-03-17 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Anemia
Keywords: APG-5918; Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Ascending Dose (SAD) cohorts in Healthy Subjects (Part A) (Experimental): Subjects will be randomized to receive a single dose of APG-5918 or placebo.
  Interventions: Drug: APG-5918; Drug: Placebo
- Multiple Ascending Dose (MAD) cohorts in Anemic Patients (Part B) (Experimental): Subjects will receive once daily APG-5918 for 84 days or till EOT.
  Interventions: Drug: APG-5918

INTERVENTIONS:
Drug: APG-5918 — oral tablets 10mg, 50mg, 200mg.
Drug: Placebo — Matching placebo
  Arms: Single Ascending Dose (SAD) cohorts in Healthy Subjects (Part A)

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, pharmacokinetics and efficacy of APG-5918 in Healthy Subjects or Anemic Patients.

DETAILED DESCRIPTION:
The trial has two parts. Part A is a randomized, double-blind, placebo- controlled, single-dose escalation study in up to 7 cohorts to evaluate the safety, tolerability, and PK characteristics of APG-5918 in healthy subjects and to explore whether MTDS will be achieved within the range of projected therapeutic doses for anemia.

Part B is an opened-label,, multi-dose escalation trial in up to 6 cohorts to evaluate the safety, tolerability, PK and preliminary efficacy of APG-5918 in anemic subjects.

ELIGIBILITY:
Inclusion Criteria:

-

1.Inclusion criteria for healthy subjects

1. Age ≥ 18 years and ≤ 55 years.
2. Body mass index (BMI) 18~28kg/m² (inclusive).
3. Hb: 120 g/L~160 g/L (inclusive).
4. Normal iron stores (normal serum iron and serum ferritin).

2.Inclusion criteria for anemic subjects

1. Age ≥ 18 years.
2. Chronic patients with anemia, including but not limited to β-thalassemia, with Hb ≤ 100 g/L at screening.
3. BMI: 16~32 kg/m2 (inclusive).
4. Serum folate and vitamin B12 levels above lower limit of normal (LLN).
5. Ferritin ≥ 40 ng/mL.
6. ALT, AST ≤ 2 × ULN, or Direct (Unbound) total bilirubin (DBIL) ≤ 2.0× ULN.
7. No active or chronic bleeding.
8. ECOG performance status score of 0 to 1.

3. Female subjects of childbearing potential who have a negative serum or urine pregnancy test within 7 days prior to the first dose.

4. Subjects and their partners volunteer to use protocol-specified effective contraception during treatment and for at least 3 months after the last dose of study drug (see Section 8.7 for details).

5. Ability to understand and willingness to sign a written informed consent form (the consent form must be signed by the subject prior to any study-specific procedures).

Exclusion criteria

1.Exclusion criteria for healthy subjects

1. History of any disease or clinical condition that, in the opinion of the investigator, could confound the results of the study or pose an additional risk to the subject by administering study drug. Including but not limited to history or presence of cardiac, endocrine, hematologic, hepatic, gastrointestinal, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other diseases.
2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 × upper limit of normal (ULN), or total bilirubin (TBIL) > 1.5 × ULN at screening.
3. Surgery (except minor cosmetic surgery or minor dental surgery) within 3 months prior to screening.
4. Blood donation or blood loss of more than 400 ml within 3 months before screening or plans to donate blood or blood components during the study.
5. Use of another investigational product within 30 days or 5 half-lives, whichever is longer, or currently participating in a prospective study of an investigational product or medical device.
6. History of addictive substance abuse.
7. Alcohol breath test fails.

2.Exclusion criteria for anemic subjects

1. Clinically significant or uncontrolled persistent autoimmune diseases (e.g., rheumatoid arthritis, Crohn's disease, celiac disease, etc.).
2. Uncontrolled hypertension (diastolic blood pressure > 110 mmHg or systolic blood pressure > 170 mmHg at screening) or diabetes as judged by the investigator.
3. New York Heart Association Class II to IV congestive heart failure, or recent myocardial infarction or acute coronary syndrome.
4. History of diagnosis of persistent hemolysis or hemolytic syndrome except for hypoferric anemia and beta-thalassemia.
5. History of thrombosis or new blood clots within 4 weeks prior to screening.
6. Any active infection requiring systemic antibiotics within 14 days prior to the first dose administration.
7. Intravenous iron within 28 days prior to screening.
8. Previous history of organ transplantation.
9. Patients who participated in other clinical studies within 4 weeks prior to the first dose administration and were still taking other study drugs or had not exceeded 5 half-lives.

3.Positive screening results for hepatitis B virus surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus antibody (HIV Ab), or treponema pallidum antibody at screening.

4.Standard 12-lead ECG QTcB > 450 ms in men and > 470 ms in women. 5. History of regular alcohol consumption within 6 months before screening, daily average intake of ethanol ≥ 30 grams (male) or ≥ 20 grams (female).

6. Female subjects who are pregnant, planning to become pregnant, or breastfeeding, or male subjects whose partners intend to become pregnant.

7. Any subject who is not suitable for participating in this study as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-07-15 (Estimated)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Events (TEAEs) | up to 7 days in Part A and 84 days or till EOT in Part B
  TEAEs will be assessed via CTCAE version 5.0 based on the frequency of adverse events/serious adverse events (AEs/SAEs), clinically significant laboratory test results, 12-lead ECGs, and vital signs.

SECONDARY OUTCOMES:
Plasma Concentrations of APG-5918 | Days 1, 2 and 3 in Part A; Days 1, 15 and 28 in Part B
  Blood samples will be collected to measure the plasma concentration of APG-5918 by a validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) method.
Measurement of Hemoglobin | 84 days or till EOT in Part B
  Change from baseline in hemoglobin will be measured in peripheral whole blood by flow cytometry.

OTHER OUTCOMES:
Expression levels of H3K27me3 | 84 days or till EOT in Part B
  Expression levels of H3K27me3 in circulating monocytes will be evaluated by fluorescence-activated cell sorting (FACS).

CONTACTS AND LOCATIONS:
Overall Officials: Zhongyuan Xu, M.D.,Ph.D., Principal Investigator — Nanfang Hospital, Southern Medical University; Yang Liang, M.D.,Ph.D., Principal Investigator — Sun Yat-sen University
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong